CLINICAL TRIAL: NCT04839302
Title: Detection and Delineation of Necrotizing Fasciitis Via a Vascular Perfusion Fluorophore: A Pilot Study
Brief Title: Detection and Delineation of Necrotizing Fasciitis Via a Vascular Perfusion Fluorophore
Status: Completed | Type: Observational
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Principal Investigator, Eric R. Henderson, Associate Professor of Orthopaedics, Dartmouth-Hitchcock Medical Center
Other Study IDs: STUDY02000905
Record Dates: First submitted 2021-04-08; First posted 2021-04-09 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Necrotising Fasciitis
Keywords: indocyanine green; Necrotising Fascitis
MeSH Terms: conditions — Fasciitis, Necrotizing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with possible nectrotizing fascitis: Patients with clinical suspicion of necrotizing fasciitis would receive a weight-appropriate IV dose of indocyanine green (ICG, FDA-approved) with immediate fluorescence imaging of the affected body part and simultaneous imaging of an unaffected region
  Interventions: Drug: Indocyanine green solution

INTERVENTIONS:
Drug: Indocyanine green solution — Patients with clinical suspicion of necrotizing fasciitis would receive a weight-appropriate IV dose of indocyanine green (ICG, FDA-approved) with immediate fluorescence imaging of the affected body part and simultaneous imaging of an unaffected region

SUMMARY:
The primary objective of this work is to determine if fluorescence signal intensity changes from a vascular perfusion fluorophore (indocyanine green) can be associated with the presence of necrotizing fasciitis.

Hypothesis - Tissue regions affected with necrotizing fasciitis will demonstrate reduced fluorescence intensity compared to an unaffected region without clinical evidence of necrotizing fasciitis.

DETAILED DESCRIPTION:
Necrotizing fasciitis (NF)-commonly known as 'flesh-eating bacteria'-is an aggressive soft-tissue infection that has a high mortality rate (30-50%). NF is generally associated with traumatic inoculation of extremely aggressive bacteria into the soft-tissues surrounding the fascial layer of connective tissue, just deep to the subcutaneous fat. This tissue layer provides an ideal environment for bacterial growth and also facilitates rapid advancement of the bacteria along the fascia. The result is a soft-tissue infection that often spreads centrally prior to detection and/or adequate management, leading to systemic sepsis, multi-organ failure, and death.

Further complicating NF management is that there is no definitive diagnostic test. Patients with NF present generally with pain, fever, and elevated inflammatory labs (white blood cell count (WBC), erythrocyte sedimentation rate (ESR), and C-reactive protein (CRP)), other lab abnormalities (elevated glucose and creatinine; reduced sodium and hemoglobin); however, these are non-specific findings that are associated with numerous other-nonfatal-conditions. For this reason, a diagnosis of NF is often missed until the condition has progressed too far.

Medical fluorescence is a nascent form of medical imaging that seeks to improve the recognition of important anatomical structures and disease processes through machine-assisted, visual identification using fluorescent probes called fluorophores. Several types of fluorophores exist: targeted fluorophores, enzyme-activated fluorophores, and simple intravascular fluorophores.

Intravascular fluorophores, primarily indocyanine green (ICG), have been available for ~100 years. ICG is FDA approved and has an excellent safety record with no demonstrable toxicity. When injected intravenously and viewed with an appropriate fluorescence imager, ICG effectively maps out the local vasculature, enabling the viewer to distinguish perfused and non-perfused tissues. ICG's FDA-approved indications and uses include angiography to determine cardiac output, hepatic function, liver blood flow, and ophthalmic anatomy.

Upon histological examination of tissues affected by NF, there exist four commonly observed features: 1) the presence of bacteria; 2) robust neutrophil infiltration; 3) tissue necrosis; 4) vascular thrombosis. DH-H Department of Pathology currently reviews tissue biopsies with respect to these criteria when evaluating tissue for the presence of necrotizing fasciitis (Soloman et al, Modern Pathology, 2018, pp 546-552). While useful to guide clinical decision-making, histological review is not considered to be a definitive diagnostic finding, but these observations do have moderate sensitivity and specificity with culture data, which is considered to be the ultimate determinant of an NF diagnosis.

Because of the profound pro-thrombotic effects of necrotizing fasciitis within the subcutaneous tissues, we hypothesize that the administration of ICG and subsequent imaging of a bodily region affected with NF will demonstrate substantially reduced fluorescence compared to the patient's unaffected tissues. If we can demonstrate that ICG fluorescence voids are characteristic of NF, this could potentially lead to a more rapid, and potentially more accurate, diagnosis of NF that would lead to more rapid definitive management and-likely-improved outcomes.

The goal of this pilot study is to evaluate whether ICG fluorescence may be used as a non-invasive method of identifying the presence of NF.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older
2. Clinical suspicion of necrotizing fasciitis based on physician or mid-level provider assessment. Clinical suspicion would be based upon the presence of one or more of these findings: Pain out of proportion to visible findings Temperature 100.4 F LRINEC (Laboratory Risk INdicator for NECrotizing fasciitis) score of ≥6 (https://pubmed.ncbi.nlm.nih.gov/15241098/) Tense soft tissues
3. Determined to be a candidate for soft-tissue biopsy and/or surgical debridement by the on-call emergency department, orthopaedic, and/or general surgical trauma teams.
4. The ability to give written informed consent

Exclusion Criteria:

1. History of allergy to ICG and/or iodine
2. Pregnant women or nursing mothers
3. No comparator region available for imaging control

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects presenting to the Emergency Department (ED) with clinical suspicion for necrotizing fasciitis (history, exam, lab studies, imaging studies).
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2021-04-05 (Actual); Primary Completion 2024-12-04 (Actual); Study Completion 2024-12-04 (Actual)

PRIMARY OUTCOMES:
Diagnosis of Necrotising Fascitis using indocyanine green | One Day
  Administration of ICG and subsequent imaging of a bodily region affected with NF will demonstrate substantially reduced fluorescence compared to the patient's unaffected tissues. Demonstration that ICG fluorescence voids are characteristic of NF.

CONTACTS AND LOCATIONS:
Overall Officials: Eric R Henderson, MD, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Dartmouth-Hitchock, Lebanon, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Solomon IH, Borscheid R, Laga AC, Askari R, Granter SR. Frozen sections are unreliable for the diagnosis of necrotizing soft tissue infections. Mod Pathol. 2018 Apr;31(4):546-552. doi: 10.1038/modpathol.2017.173. Epub 2017 Dec 15. PMID 29243739
- [Background] Betz CS, Zhorzel S, Schachenmayr H, Stepp H, Havel M, Siedek V, Leunig A, Matthias C, Hopper C, Harreus U. Endoscopic measurements of free-flap perfusion in the head and neck region using red-excited Indocyanine Green: preliminary results. J Plast Reconstr Aesthet Surg. 2009 Dec;62(12):1602-8. doi: 10.1016/j.bjps.2008.07.042. Epub 2008 Nov 25. PMID 19036663
- [Derived] Ray GS, Streeter SS, Bateman LM, Elliott JT, Henderson ER; NEFARIOUS Study Group. Real-time identification of life-threatening necrotizing soft-tissue infections using indocyanine green fluorescence imaging. J Biomed Opt. 2024 Jun;29(6):066003. doi: 10.1117/1.JBO.29.6.066003. Epub 2024 May 14. PMID 38745983